CLINICAL TRIAL: NCT04771312
Title: Online Network Intervention to Increase HIV Pre-exposure Prophylaxis Intention: A Mobile App-based Experiment
Brief Title: Online Network Intervention to Increase HIV Pre-exposure Prophylaxis Intention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1707085
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Behavior, Health
Keywords: PrEP; HIV prevention
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Information-only intervention (Active Comparator): Participants are randomly assigned to 6-person peer networks in a mobile app. Participants in the information-only condition could respond to daily questions in a diary.
  Interventions: Behavioral: Mobile app information-only intervention
- Social support network intervention (Experimental): Participants are randomly assigned to 6-person peer networks in a mobile app. Participants in the social support condition could use an online chatting tool where they can send messages to their own network.
  Interventions: Behavioral: Mobile app social support network intervention

INTERVENTIONS:
Behavioral: Mobile app information-only intervention — Mobile app intervention. Participants view information regarding PrEP that address beliefs and barriers surrounding adoption and uptake. Participants can respond to daily questions in a diary. Participants can also use a locator tool to find where PrEP can be found near them.
  Arms: Information-only intervention
Behavioral: Mobile app social support network intervention — Mobile app intervention. Participants view information regarding PrEP that address beliefs and barriers surrounding adoption and uptake. Participants are shown an online chatting tool where they can discuss with each other and answer daily questions. Participants can also use a locator tool to find where PrEP can be found near them.
  Arms: Social support network intervention

SUMMARY:
HIV pre-exposure prophylaxis (or PrEP) is an effective additional preventative measure for reducing the risk of HIV transmission. To address low levels of uptake, there is a need for public health interventions to increase target populations' awareness and willingness for adopting PrEP. One potential solution may be to incorporate a network intervention, which utilizes the connections between individuals to facilitate health behavior. This project examines how online networks can influence PrEP adoption intentions among gay and bisexual men through a mobile app-based experiment. In this study, participants will be randomly assigned into a social support condition or information-only control. Both conditions will involve an information component consisting messages aimed to address awareness, knowledge, and perceived barriers of PrEP adoption. However, those in the social support condition will also have an online chatting tool where they can discuss topics surrounding PrEP.

The primary objective of this study is to test the effectiveness of the mobile app intervention in increasing participants' knowledge/attitudes/intentions to initiate PrEP.

The secondary objective of this study is to determine the mechanism of the intervention through mediation analyses.

DETAILED DESCRIPTION:
Roughly 1.7 million people worldwide are infected with HIV each year (UNAIDS, 2017). HIV pre-exposure prophylaxis (or PrEP) refers to taking a daily oral medicine to reduce the risk of contracting HIV. Known by the brand name Truvada or Descovy, PrEP is an effective additional preventative measure for reducing the risk of HIV transmission. To address low levels of uptake, there is a need for public health interventions to increase target populations' awareness and willingness for adopting PrEP.

One potential solution may be to incorporate a network intervention, which utilizes the connections between individuals to facilitate health behavior. In particular, online networks can provide anonymous support that transcends geographical boundaries (DeAndrea, 2015). Stigmatized behaviors, such as the adoption of PrEP, may greatly benefit from interventions that utilize online networks. This project examines how online networks can influence PrEP adoption intentions among gay and bisexual men through a mobile app-based experiment.

There are several ways in which online networks may influence health; however, social support may serve as the primary mechanism that influences PrEP adoption. In the context of HIV prevention, social support has generally reduced HIV-related risky behaviors (Qiao, Li, & Stanton, 2014). Thus, it is important to consider social support as a factor than can influence one's intention to adopt PrEP.

This field experiment will randomly assign participants into a social support condition or information-only control, and then randomly assign them into homophilous, clustered six-member peer networks. Both conditions will involve an information component consisting messages aimed to address awareness, knowledge, and perceived barriers of PrEP adoption. Social support will be operationalized through an online chatting tool where participants can discuss topics surrounding PrEP.

The primary objective of this study is to test the effectiveness of the mobile app intervention in increasing participants' knowledge/attitudes/intentions to initiate PrEP.

The secondary objective of this study is to determine the mechanism of the intervention through mediation analyses.

ELIGIBILITY:
Inclusion Criteria:

* Gay or bisexual male
* Aged 18 and 35
* HIV-negative
* Not on PrEP
* Using an Android smartphone

Exclusion Criteria:

* Already participating in another HIV-related study.
* Not able or willing to carry an Android smartphone.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Must identify as male and be assigned male at birth.
Enrollment: 50 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Intention to start PrEP | Baseline and 1 week
  3-item measure based on the Reasoned Action Approach for intention to start PrEP from 1 = "strongly disagree" to 5 = "strongly agree."
Change from baseline on Attitude toward starting PrEP | Baseline and 1 week
  7-point semantic differential measure based on the Reasoned Action Approach for attitude to start PrEP with items such as "Good/Bad" and "Useful/Useless."
Change from baseline on Knowledge of PrEP | Baseline and 1 week
  4-items on functional knowledge of HIV pre-exposure prophylaxis. Options include "True," "False," and "Unsure."

SECONDARY OUTCOMES:
Perceived Social Support | 1 week
  Validated measure of perceived informational and emotional support from 1 = "strongly disagree" to 5 = "strongly agree."

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers.